CLINICAL TRIAL: NCT03432130
Title: The Effect of Structured Training Program and Body Composition on Injury Occurrence in Hip-hop Dance
Brief Title: Injury Occurrence in Hip-hop Dance
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Ljubljana (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Prevention
Other Study IDs: HIP-HOP INJURIES
Record Dates: First submitted 2018-02-07; First posted 2018-02-14 (Actual); Last update posted 2019-04-24 (Actual); Status verified 2019-04

CONDITIONS: Sports Injury; Body Composition
Keywords: hip-hop dance, injuries, body fat
MeSH Terms: conditions — Athletic Injuries; Wounds and Injuries

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Experimental group (Experimental): Performing a structural training program twice a week, 30 minutes each.
  Interventions: Other: Structural training program
- Control group (No Intervention)

INTERVENTIONS:
Other: Structural training program — 15-week experimental structural training protocol
  Arms: Experimental group

SUMMARY:
The study will investigate the effect of structural training program and body composition on injury occurrence in hip-hop dance. Assuming that training program can significantly lower the number of injuries (experimental group will have less injuries during and at the end of the trial) and that body fat percentage negatively effects injury occurrence (dancers with higher body fat percentage will be more often injured).

ELIGIBILITY:
Inclusion Criteria:

* hip-hop dancer (active)

Exclusion Criteria:

* injured

Min Age: 14 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Enrollment: 100 (Actual)
Dates: Start 2017-09-30 (Actual); Primary Completion 2018-06-30 (Actual); Study Completion 2018-09-30 (Actual)

PRIMARY OUTCOMES:
Number of injuries | 3 months

CONTACTS AND LOCATIONS:
Locations (1):
- University of Ljubljana, Faculty of Sport, Ljubljana, Slovenia

IPD SHARING:
Plan to Share IPD: Undecided